CLINICAL TRIAL: NCT00818597
Title: PhaseI/II Study of the Safety and Efficacy of the Use of Granulocyte-Concentrates Applied in Extracorporeal Circulation Devices-the EISS-1 Study
Brief Title: Extracorporeal Immune Support System (EISS) for the Treatment of Septic Patients
Acronym: EISS-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rostock (Other)
Responsible Party: Steffen Mitzner/ Head Division of Nephrology, University of Rostock, Medical Faculty
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EISS-1
Record Dates: First submitted 2009-01-05; First posted 2009-01-07 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Severe Sepsis and Septic Shock
Keywords: septic shock; immunoparalysis; extracorporeal; granulocyte bioreactor; plasmapheresis
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EISS-treatment (Experimental): In this arm patients receive additional treatment with the EISS-bioreactor
  Interventions: Device: EISS

INTERVENTIONS:
Device: EISS — Two six hour-treatments with the EISS-Immune-cell bioreactor device within 72 hours post inclusion.

SUMMARY:
The purpose of this study is to investigate the effect of an extracorporeal application of a bed-side bioreactor containing human donor granulocytes on the course and outcome of septic shock in humans.

ELIGIBILITY:
Inclusion Criteria:

* sepsis with at least one organ failure (severe sepsis) or septic shock

Exclusion Criteria:

* Participation in another study within the last 30 days
* Earlier participation in this study
* Pregnancy
* Bleeding, clinically not controlled (needing more than 2 red blood cell-transfusions per day)
* Hemodynamic shock for more than 12 hours (systolic BP <90mmHg) despite adequate therapy
* HIV infection
* HCV infection, active

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-12; Primary Completion 2004-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
single organ functions (circulation, kidney, lung, liver) | 28day post inclusion

SECONDARY OUTCOMES:
survival | 28day post inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rostock, Department of Medicine, Division of Nephrology, Rostock, Germany

REFERENCES:
- [Background] Mitzner SR, Freytag J, Sauer M, Kleinfeldt T, Altrichter J, Klohr S, Koball S, Stange J, Ringel B, Nebe B, Schmidt H, Podbielski A, Noeldge-Schomburg G, Schmidt R. Use of human preconditioned phagocytes for extracorporeal immune support: introduction of a concept. Ther Apher. 2001 Oct;5(5):423-32. doi: 10.1046/j.1526-0968.2001.00378.x. PMID 11778929
- [Background] Sauer M, Altrichter J, Kreutzer HJ, Logters T, Scholz M, Noldge-Schomburg G, Schmidt R, Mitzner SR. Extracorporeal cell therapy with granulocytes in a pig model of Gram-positive sepsis. Crit Care Med. 2009 Feb;37(2):606-13. doi: 10.1097/CCM.0b013e318194aa77. PMID 19114920
- [Derived] Altrichter J, Sauer M, Kaftan K, Birken T, Gloger D, Gloger M, Henschel J, Hickstein H, Klar E, Koball S, Pertschy A, Noldge-Schomburg G, Vagts DA, Mitzner SR. Extracorporeal cell therapy of septic shock patients with donor granulocytes: a pilot study. Crit Care. 2011;15(2):R82. doi: 10.1186/cc10076. Epub 2011 Mar 3. PMID 21371308